CLINICAL TRIAL: NCT00291031
Title: A Randomised Controlled Trial of Imagery Rehearsal Therapy (IRT) of Nightmares in a Psychiatric Population
Brief Title: Study of the Effect of Imagery Rehearsal Therapy (IRT) of Nightmares
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GGZ Centraal (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Principal Investigator, Annette van Schagen, Clinical psychologist, GGZ Centraal
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WO-SG-114NM
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Nightmares; Anxiety Disorders; Mood Disorders; Personality Disorders
Keywords: nightmare; sleep disorder; sleep; imagery rehearsal; anxiety disorders; mood disorders; personality disorders
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Personality Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IRT (Experimental): Patients randomly assigned to the IRT condition receive Imagery Rehearsal Therapy after 4 weeks since the entrance into the trial next to their treatment as usual.
  Interventions: Behavioral: Imagery Rehearsal Therapy (IRT)
- TAU (No Intervention): Patients that are randomly assigned to the waiting list control condition get treatment as usual (TAU) and complete the daily nightmare logs for a period of three months. These patients get the IRT intervention after waiting for 6 months.

INTERVENTIONS:
Behavioral: Imagery Rehearsal Therapy (IRT) — Imagery Rehearsal Therapy is given by psychologists, psychotherapists or psychiatrists. The IRT therapists are all trained by Annette van Schagen, principal investigator.
  IRT consists of six 1-hour sessions. The six sessions are given in a period of three months. Each session is described in the IRT Manual. The IRT Manual is devised by the principal investigator Annette van Schagen in colaboration with Victor Spoormaker PhD. There is a patient version of the IRT manual available for the patients, which includes descriptions of the IRT sessions and homework assignments.
  Other Names: IRT
  Arms: IRT

SUMMARY:
The purpose of this study is to determine whether Imagery Rehearsal Therapy(IRT) is effective in the reduction of the number of nightmares and the nightmare distress in a population of patients with psychiatric disorders.

DETAILED DESCRIPTION:
Within the normal population 4-8% of the people suffer regularly from nightmares. Clinical observations show that nightmares are a common problem for patients who suffer from all kinds of psychiatric disorders, and not just for the patients diagnosed with PTSD. Often nightmares can lead to sleep disorders, which have a negative impact on emotional well-being and cognitive functioning during the day. As well as this a strong relationship between severity of nightmares and severity of psychopathology has been found. This gives a strong argument for treatment of nightmares as a symptom, separate from the psychiatric disorder.

A few controlled studies of the treatment of nightmares have been published, in which behavioral therapy, relaxation techniques, exposure and systematic desensitization have been studied, all of which have shown positive results. But these techniques do not seem to reduce the number of nightmares in patients who suffer from PTSD. These last few years more controlled studies of a cognitive behavioral technique called 'Imagery Rehearsal Therapy' (IRT) have been published. With IRT patients have to change the script of their nightmares into a different outcome, and rehearse this new script using cognitive imagery a few times a day.

Comparisons: treatment of nightmares with IRT compared to a waitlist control group who do not get IRT until 6 months later.

ELIGIBILITY:
Patients referred to GGZ Centraal (previously Symfora groep) by their family doctor/GP for treatment of a psychiatric disorder. Patients that suffer from anxiety disorders, eating disorders, mood disorders and/or personality disorders.

Inclusion Criteria:

* Minimum of 3 nightmares per month
* Nightmares are associated with distress in daily life
* Subject wants to get treatment for the nightmares

Exclusion Criteria:

* Imagery rehearsal therapy for nightmares in the past
* Psychotic disorders
* Acute psychiatric crisis
* Mentally challenged or neuropsychiatric syndrome
* Severe addiction problems
* Insufficient mastery of the Dutch language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-02; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Frequency of nightmares scored in prospective daily nightmare logs | Daily logs for 18 weeks, then periods of 4 weeks every 3 months
Frequency of nightmares scored on the Nightmare Frequency Questionnaire | At beginning of trial, 4, 16, 30, 42 and 56 weeks

SECONDARY OUTCOMES:
Intensity of nightmares scored in prospective daily nightmare logs | Daily logs for 18 weeks, then periods of 4 weeks every 3 months
Effects of nightmares scored on the Nightmare Effects Survey | 1, 4, 16, 30, 42 and 56 weeks
Nightmare distress scored on the Nightmare Distress Questionnaire | 1, 4, 16, 30, 42 and 56 weeks
Sleep problems scored on the SLEEP-50 | 1, 4, 16, 30, 42 and 56 weeks
Psychiatric symptoms scored on the Symptom Check List (SCL-90) | 1, 4, 16, 30, 42 and 56 weeks
Symptoms of post-traumatic stress disorder scored on the Zelf Inventarisatie Lijst PTSS ZIL (= PTSD Inventory) | 1, 4, 16, 30, 42 and 56 weeks
Quality of life scored on the abbreviated World Health Organization Quality of Life scale (WHOQoL-Bref) | 1, 4, 16, 30, 42 and 56 weeks
Nightmare efficacy and content measured by Nightmare Efficacy & Content Questionnaire | 1, 4, 16, 30, 42 and 56 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Annette M. van Schagen, MA, Principal Investigator — GGZ Centraal (previously Symfora groep); Jan van den Bout, PhD, Study Chair — Utrecht University; Victor I. Spoormaker, PhD, Study Chair — Max-Planck-Institute of Psychiatry; Jaap Lancee, PhD, Study Chair — University of Amsterdam
Locations (3):
- Netherlands (3):
  - GGZ Centraal, De Meregaard, Almere Stad
  - GGZ Centraal, Zon & Schild, Amersfoort
  - GGZ Centraal, De Rembrandthof, Hilversum

REFERENCES:
- [Background] Krakow B, Hollifield M, Johnston L, Koss M, Schrader R, Warner TD, Tandberg D, Lauriello J, McBride L, Cutchen L, Cheng D, Emmons S, Germain A, Melendrez D, Sandoval D, Prince H. Imagery rehearsal therapy for chronic nightmares in sexual assault survivors with posttraumatic stress disorder: a randomized controlled trial. JAMA. 2001 Aug 1;286(5):537-45. doi: 10.1001/jama.286.5.537. PMID 11476655
- [Background] Spoormaker VI, Schredl M, van den Bout J. Nightmares: from anxiety symptom to sleep disorder. Sleep Med Rev. 2006 Feb;10(1):19-31. doi: 10.1016/j.smrv.2005.06.001. Epub 2005 Dec 27. PMID 16377217
- [Background] Benca RM, Obermeyer WH, Thisted RA, Gillin JC. Sleep and psychiatric disorders. A meta-analysis. Arch Gen Psychiatry. 1992 Aug;49(8):651-68; discussion 669-70. doi: 10.1001/archpsyc.1992.01820080059010. PMID 1386215
- [Background] Blagrove M, Farmer L, Williams E. The relationship of nightmare frequency and nightmare distress to well-being. J Sleep Res. 2004 Jun;13(2):129-36. doi: 10.1111/j.1365-2869.2004.00394.x. PMID 15175092
- [Background] Rothbaum BO, Mellman TA. Dreams and exposure therapy in PTSD. J Trauma Stress. 2001 Jul;14(3):481-90. doi: 10.1023/A:1011104521887. PMID 11534880
- [Background] Spoormaker VI, Verbeek I, van den Bout J, Klip EC. Initial validation of the SLEEP-50 questionnaire. Behav Sleep Med. 2005;3(4):227-46. doi: 10.1207/s15402010bsm0304_4. PMID 16190812
- [Background] Strine TW, Chapman DP. Associations of frequent sleep insufficiency with health-related quality of life and health behaviors. Sleep Med. 2005 Jan;6(1):23-7. doi: 10.1016/j.sleep.2004.06.003. PMID 15680291
- [Background] van de Willige G, Wiersma D, Nienhuis FJ, Jenner JA. Changes in quality of life in chronic psychiatric patients: a comparison between EuroQol (EQ-5D) and WHOQoL. Qual Life Res. 2005 Mar;14(2):441-51. doi: 10.1007/s11136-004-0689-y. PMID 15892433
- [Derived] van Schagen AM, Lancee J, de Groot IW, Spoormaker VI, van den Bout J. Imagery rehearsal therapy in addition to treatment as usual for patients with diverse psychiatric diagnoses suffering from nightmares: a randomized controlled trial. J Clin Psychiatry. 2015 Sep;76(9):e1105-13. doi: 10.4088/JCP.14m09216. PMID 26455674
- See also: A website with information on nightmares, and other sleep problems. Sponsored by Utrecht University and Fonds Psychische Gezondheid — http://www.nachtmerries.org/
- See also: The website of Symfora groep, Centres for Mental Health Care — http://www.symfora.nl